CLINICAL TRIAL: NCT02992548
Title: Effect of Pravastatin on Erythrocyte Membrane Fatty Acid Contents in Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, WON SUK AN, Professor, Dong-A University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: prava_2016
Record Dates: First submitted 2016-12-10; First posted 2016-12-14 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; pravastatin; erythrocyte membrane fatty acid
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pravastatin group (Experimental): Use of pravastatin 20mg to 40mg
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin

SUMMARY:
Treatment using statin has been decreased the risk of cardiovascular events in pre-dialysis CKD population. Supplementation with omega-3 fatty acid (FA) lowers the risk of cardiovascular death in patients with myocardial infarction. This cardioprotective effect of omega-3 FA can be explained by anti-inflammatory, anti-oxidative, or anti-thrombotic effects. Statin such as pravastatin is also known to have anti-inflammatory and antioxidant properties, suggesting that statin may replace the cardioprotective effect of omega-3 fatty acids. Erythrocyte membrane oleic acid is significantly higher in patients with acute coronary syndrome than control subjects. The cardioprotective effect of omega-3 FA may also be related to decreased oleic acid content of erythrocyte membrane. There is no report about the effect of statin on FA including erythrocyte membrane oleic acid. As omega-3 FAs are recognized as therapeutic agents for reducing triglycerides, statin may affect on the erythrocyte membrane FA. Therefore, pravastatin supplementation can modify erythrocyte membrane FA contents including oleic acid in CKD patients.

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) have higher risk of death and cardiovascular disease than general population. Treatment using statin has been decreased the risk of cardiovascular events in pre-dialysis CKD population. Supplementation with omega-3 fatty acid (FA) lowers the risk of cardiovascular death in patients with myocardial infarction. This cardioprotective effect of omega-3 FA can be explained by anti-inflammatory, anti-oxidative, or anti-thrombotic effects. Statin such as pravastatin is also known to have anti-inflammatory and antioxidant properties, suggesting that statin may replace the cardioprotective effect of omega-3 fatty acids.

Omega-3 FA such as EPA (eicosapentaenoic acid), DHA (docosahexaenoic acid), and EPA/arachidonic acid ratio are well known as key indicators of cardiovascular disease. In addition, erythrocyte membrane oleic acid is significantly higher in patients with acute coronary syndrome than control subjects. The cardioprotective effect of omega-3 FA may also be related to decreased oleic acid content of erythrocyte membrane. There is no report about the effect of statin on FA including erythrocyte membrane oleic acid. As omega-3 FAs are recognized as therapeutic agents for reducing triglycerides, statin may affect on the erythrocyte membrane FA. Therefore, pravastatin supplementation can modify erythrocyte membrane FA contents including oleic acid in CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients who agreed with written informed consent
* CKD patients who do not take statin
* Who have LDL cholesterol over 100mg/dL and coronary vascular disease(CVD) or equivalent risk; Who have LDL cholesterol over 130mg/dL and two or more coronary vascular risk; Whose LDL cholesterol over 160mg/dL in patient with CKD stage 1 to 5 without dialysis.

Exclusion Criteria:

* Patients with acute illness, a history of active infection, CVD, acute kidney injury during the past 3 months, or a history of malignancy or liver disease
* Patients using statin, omega-3 fatty acid or sevelamer hydrochloride within 3 months
* Patients who experienced side effects by statin treatment
* Pregnant or pregnancy expected CKD patients
* Patient with dyslipidemia due to nephrotic syndrome
* Patient taken imaging study using contrast media during the past 14 days
* Patient with albumin level < 3.0 g/dL

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-09; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
mean change of erythrocyte membrane fatty acid including oleic acid | 24 weeks after intervention

SECONDARY OUTCOMES:
mean change of total cholesterol | 24 weeks after intervention
mean change of triglyceride | 24 weeks after intervention
mean change of LDL-cholesterol | 24 weeks after intervention
mean change of HDL-cholesterol | 24 weeks after intervention
mean change of adiponectin | 24 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Won Suk An, MD, Principal Investigator — Dong-A University; Yeong Hoon Kim, MD, Study Director — Inje University
Locations (2):
- South Korea (2):
  - Dong-A University, Busan
  - Inje University, Pusan Paik Hospital, Busan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tonelli M, Muntner P, Lloyd A, Manns B, Klarenbach S, Pannu N, James M, Hemmelgarn B; Alberta Kidney Disease Network. Association between LDL-C and risk of myocardial infarction in CKD. J Am Soc Nephrol. 2013 May;24(6):979-86. doi: 10.1681/ASN.2012080870. Epub 2013 May 16. PMID 23687359
- [Background] Tonelli M, Muntner P, Lloyd A, Manns BJ, Klarenbach S, Pannu N, James MT, Hemmelgarn BR; Alberta Kidney Disease Network. Risk of coronary events in people with chronic kidney disease compared with those with diabetes: a population-level cohort study. Lancet. 2012 Sep 1;380(9844):807-14. doi: 10.1016/S0140-6736(12)60572-8. Epub 2012 Jun 19. PMID 22717317
- [Background] Stenvinkel P, Heimburger O, Paultre F, Diczfalusy U, Wang T, Berglund L, Jogestrand T. Strong association between malnutrition, inflammation, and atherosclerosis in chronic renal failure. Kidney Int. 1999 May;55(5):1899-911. doi: 10.1046/j.1523-1755.1999.00422.x. PMID 10231453
- [Background] Baigent C, Landray MJ, Reith C, Emberson J, Wheeler DC, Tomson C, Wanner C, Krane V, Cass A, Craig J, Neal B, Jiang L, Hooi LS, Levin A, Agodoa L, Gaziano M, Kasiske B, Walker R, Massy ZA, Feldt-Rasmussen B, Krairittichai U, Ophascharoensuk V, Fellstrom B, Holdaas H, Tesar V, Wiecek A, Grobbee D, de Zeeuw D, Gronhagen-Riska C, Dasgupta T, Lewis D, Herrington W, Mafham M, Majoni W, Wallendszus K, Grimm R, Pedersen T, Tobert J, Armitage J, Baxter A, Bray C, Chen Y, Chen Z, Hill M, Knott C, Parish S, Simpson D, Sleight P, Young A, Collins R; SHARP Investigators. The effects of lowering LDL cholesterol with simvastatin plus ezetimibe in patients with chronic kidney disease (Study of Heart and Renal Protection): a randomised placebo-controlled trial. Lancet. 2011 Jun 25;377(9784):2181-92. doi: 10.1016/S0140-6736(11)60739-3. Epub 2011 Jun 12. PMID 21663949
- [Background] Wanner C, Tonelli M; Kidney Disease: Improving Global Outcomes Lipid Guideline Development Work Group Members. KDIGO Clinical Practice Guideline for Lipid Management in CKD: summary of recommendation statements and clinical approach to the patient. Kidney Int. 2014 Jun;85(6):1303-9. doi: 10.1038/ki.2014.31. Epub 2014 Feb 19. PMID 24552851
- [Background] AIM-HIGH Investigators; Boden WE, Probstfield JL, Anderson T, Chaitman BR, Desvignes-Nickens P, Koprowicz K, McBride R, Teo K, Weintraub W. Niacin in patients with low HDL cholesterol levels receiving intensive statin therapy. N Engl J Med. 2011 Dec 15;365(24):2255-67. doi: 10.1056/NEJMoa1107579. Epub 2011 Nov 15. PMID 22085343
- [Background] Ridker PM, Pradhan A, MacFadyen JG, Libby P, Glynn RJ. Cardiovascular benefits and diabetes risks of statin therapy in primary prevention: an analysis from the JUPITER trial. Lancet. 2012 Aug 11;380(9841):565-71. doi: 10.1016/S0140-6736(12)61190-8. PMID 22883507
- [Background] Leaf A, Kang JX, Xiao YF, Billman GE. Clinical prevention of sudden cardiac death by n-3 polyunsaturated fatty acids and mechanism of prevention of arrhythmias by n-3 fish oils. Circulation. 2003 Jun 3;107(21):2646-52. doi: 10.1161/01.CIR.0000069566.78305.33. No abstract available. PMID 12782616
- [Background] Harris WS, Von Schacky C. The Omega-3 Index: a new risk factor for death from coronary heart disease? Prev Med. 2004 Jul;39(1):212-20. doi: 10.1016/j.ypmed.2004.02.030. PMID 15208005
- [Background] Block RC, Harris WS, Reid KJ, Spertus JA. Omega-6 and trans fatty acids in blood cell membranes: a risk factor for acute coronary syndromes? Am Heart J. 2008 Dec;156(6):1117-23. doi: 10.1016/j.ahj.2008.07.014. Epub 2008 Oct 14. PMID 19033007
- [Background] An WS, Kim SE, Kim KH, Lee S, Park Y, Kim HJ, Vaziri ND. Comparison of fatty acid contents of erythrocyte membrane in hemodialysis and peritoneal dialysis patients. J Ren Nutr. 2009 Jul;19(4):267-74. doi: 10.1053/j.jrn.2009.01.027. PMID 19539181
- [Background] An WS, Lee SM, Son YK, Kim SE, Kim KH, Han JY, Bae HR, Rha SH, Park Y. Omega-3 fatty acid supplementation increases 1,25-dihydroxyvitamin D and fetuin-A levels in dialysis patients. Nutr Res. 2012 Jul;32(7):495-502. doi: 10.1016/j.nutres.2012.06.005. Epub 2012 Jul 20. PMID 22901557